CLINICAL TRIAL: NCT02479919
Title: Treating Social Cognition Impairments in Patients With Schizophrenia With Repetitive Transcranial Magnetic Stimulation (Theta-Burst; TBS); a Multicentric Study
Brief Title: Treating Social Cognition With Theta Burst Stimulation: a Multicentric Study
Acronym: TBS-COG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: University Hospital, Rouen (Other); Centre Hospitalier Universitaire Dijon (Other); Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-A00424-45
Record Dates: First submitted 2015-06-02; First posted 2015-06-24 (Estimated); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Social Cognition in Patients With Schizophrenia
Keywords: theta burst stimulation; Social Cognition; Schizophrenia; transcranial magnetic stimulation
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TBS-MPC (Experimental): Intervention with Magstim® Active TBS aiming Medial Prefrontal Cortex in 18 patients with schizophrenia
  Interventions: Device: Magstim® Active TBS
- TBS-CPDLF (Active Comparator): Intervention with Magstim® Active TBS aiming Dorsolateral Prefrontal Cortex in 18 patients with schizophrenia
  Interventions: Device: Magstim® Active TBS
- TBS-Sham (Sham Comparator): Intervention with Magstim® Sham TBS in 25 patients with schizophrenia
  Interventions: Device: Magstim® Sham TBS

INTERVENTIONS:
Device: Magstim® Active TBS — Non-invasive transcranial magnetic stimulation inducing changes in cortical excitability depending on the cortical target (except for sham stimulation)
  Arms: TBS-CPDLF; TBS-MPC
Device: Magstim® Sham TBS — Sham stimulation
  Arms: TBS-Sham

SUMMARY:
The purpose of the study is to test a new treatment of social cognition deficits in patients with schizophrenia or schizoaffective disorder by transcranial magnetic stimulation (theta-burst). The study will also identify clinical, psychomotor and cognitive variables that are the most sensitive to treatment, and estimate the most sensitive treatment target between patients.

DETAILED DESCRIPTION:
The language understanding of other people is based on linguistic decoding mechanisms (phonological, semantic, syntactic ...) but also more on subtle mechanisms for the recognition of emotions and intentions. Interact with another one requires understanding its language but also to infer emotions and intentions. There are patients with schizophrenia suffering from social cognition disorders that impair social interactions; These patients often have difficulty in extracting the non-verbal emotional content of language and have difficulty inferring the thoughts and intentions of others. Recently, investigators have suggested a link between such deficits and the hypofunction of the medial prefrontal cortex.

Transcranial magnetic stimulation is a noninvasive neuromodulation technique that increases or decreases the focal cortical excitability depending on stimulation parameters. This technique is now commonly used as a therapeutic tool. It has been tried with some success in patients with schizophrenia in some indications:

* To reduce the auditory verbal hallucinations stimulating the temporal cortex
* More rarely, to reduce the negative symptoms stimulating the dorsolateral prefrontal cortex.

So far, the medial prefrontal cortex was not considered as a possible target as the scalp to cortex distance prevent from using conventional stimulation coils. Recently new coils have been developed that permit stimulation of deeper cortical regions.

Investigators hypothesize that the use of transcranial magnetic stimulation with a theta burst intermittent protocol known to increase the cortical excitability and aiming the medial prefrontal cortex with a special antenna will improve social interaction capabilities of schizophrenic patients.

In this multicentric study, involving 61 patients, investigators plan to assess the social cognition deficits before and after 10 sessions of magnetic stimulation (2 sessions per day for 5 consecutive days) using a neuronavigation system and Magstim® stimulator. In order to assess the specificity of the stimulation of medial prefrontal cortex (MPC), the effects of this treatment will be compared to the effects of the same treatment aiming the dorsolateral prefrontal cortex (DLPFC), also involved in aspects of negative symptoms of schizophrenia, and placebo effects induced by sham stimulation (using a sham coil). An anatomical MRI will be performed before the treatment to define the targets. Moreover, changes motor activity will be observed after stimulation thanks to continuous actimetry recording.

ELIGIBILITY:
Inclusion Criteria:

* with a diagnosis of schizophrenia or schizoaffective disorder (DSM-IV MINI R)
* Having signed a written informed consent
* 'Lecture Intentionnelle en situation' (LIS) score > 15 or negative 'Positive and Negative Syndrome Scale' (PANSS) score > 15

Exclusion Criteria:

* Any change in psychotropic drugs (antidepressants, antipsychotics or mood stabilizers) during the two months preceding the inclusion
* Pregnant or breastfeeding women
* Subjects with a neurological condition or with epilepsy
* Subjects with a counter-indication to MRI or Transcranial stimulation (electronic or metal implants)
* Subjects that refuse to wear earplugs during MRI

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Estimated)
Dates: Start 2017-04-11 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
V-LIS total score | change from baseline in V-LIS total score compared to 30 days after the end of the treatment

SECONDARY OUTCOMES:
Motor activity measured with an actimeter | change in baseline motor activity measured with an actimeter compared to 30 days after the end of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Dollfus, Pr, Principal Investigator — University Hospital, Caen
Locations (3):
- France (3):
  - Dollfus, Caen
  - Jaafari, Poitiers
  - Guillin, Sotteville-lès-Rouen